CLINICAL TRIAL: NCT06880965
Title: Effect of Concentrated Growth Factors on Short Implant-Supported Overdentures: a Split-Mouth Design Study.
Brief Title: Effect of Concentrated Growth Factors on Short Implant-Supported Overdentures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Atef, Lecturer at periodontology and oral medicine department Tanta university, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: R-OMPDR-8-23-2
Record Dates: First submitted 2025-03-08; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-12

CONDITIONS: Partially Edentulous Patients
Keywords: CGF, Overdenture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- short implants assisted over denture in combination with concentrated growth factors (Active Comparator): the left side of the patients' mandibular posterior region was restored with short implant in place of first molar by using short implants assisted over denture with concentrated growth factor.
  Interventions: Diagnostic Test: testing implant stability; Drug: use concentrated growth factor.; Radiation: marginal bone loss calculation
- using mandibular posterior short implants assisted over denture without concentrated growth factors (Placebo Comparator): the right side of the patients' mandibular posterior region was restored with short implant in place of first molar by using short implants assisted over denture without concentrated growth factor.
  Interventions: Diagnostic Test: testing implant stability; Radiation: marginal bone loss calculation

INTERVENTIONS:
Diagnostic Test: testing implant stability — testing implant stability by using the periotest device
Drug: use concentrated growth factor. — short implants assisted over denture in combination with concentrated growth factor.
  Arms: short implants assisted over denture in combination with concentrated growth factors
Radiation: marginal bone loss calculation — marginal bone loss calculation by digitized periapical radiograph

SUMMARY:
The purpose of this study will be to evaluate the effect of concentrated growth factors on stability and radiographic outcome of short implant supported mandibular assisted overdenture

DETAILED DESCRIPTION:
A controlled clinical trial will be performed upon patients attending the outpatient clinic of Faculty of Dentistry Tanta University.Ten male patients will be selected for this study. Split mouth study design will be used in this study where, Group I represented the right side of the patients' mandibular posterior region will be restored with short implant in place of first molar and Group II represented the left side of the patients' mandibular posterior region will be restored with short implant in place of first molar and concentrated growth factors. The patients will receive partial mandibular assisted overdenture with O-ring attachment on the implant. Stability of implant and Radiographic evaluations will be carried out for every patient at regular recall visits at the time of insertion, 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20 to 65 years old. Class I Kennedy's classification Good oral hygiene.

Exclusion Criteria:

* Bad oral hygiene. Para functional habits ex. (bruxism, clenching,)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Concentrated growth factor (CGF) Effects | one year
  evaluate the effects of concentrated growth factors on the stability of short implant-supported mandibular assisted partial overdentures. Periotest equipment was used to measure the stability of the implants in all of the patients immediately after surgery, six months later.

CONTACTS AND LOCATIONS:
Overall Officials: Sherin F Donia, PHD, Principal Investigator — Tanta University
Locations (1):
- Tanta university, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 months after puplication
Access Criteria: all the data
URL: http://www.ncbi.nlm.nih.gov/pubmed/16481614,18287085